CLINICAL TRIAL: NCT06279819
Title: Effectiveness of Gut Microbiota-targeted Dietary Intervention in Preventing Borderline Atherosclerotic Cardiovascular Disease Risk Among HIV-infected Patients
Brief Title: Effectiveness of Gut Microbiota-targeted Dietary Intervention Among HIV-infected Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junwen Yu, PhD candidate, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-008
Record Dates: First submitted 2024-01-17; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hiv; Cardiovascular Diseases; Diet, Healthy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group will receive the gut microbiota-targeted dietary intervention thrice weekly for 3 months, accompanied by bi-weekly health education videos for the same duration. The intervention will span three months, followed by a three-month follow-up period.
  Interventions: Dietary Supplement: gut microbiota-targeted dietary intervention
- control group (No Intervention): The control group will continue routine follow-up and health education practices.

INTERVENTIONS:
Dietary Supplement: gut microbiota-targeted dietary intervention — The dietary intervention used the dietary intervention plan constructed in Phase 2, on the basis of which each study participant's individual dietary habits, food preferences and economic level were taken into account.
  The dietary intervention was delivered by sending fresh ingredients. To ensure the freshness and quality of the ingredients, 2 dedicated researchers were jointly responsible for the procurement of fresh ingredients, which were purchased through regular channels on Monday, Wednesday and Friday mornings.
  Ingredients will be delivered three times a week for a 12-week intervention period. The initial food items to be sent include: 90g of fish rich in omega-3 fatty acids; 300g of vegetables and/or legumes, and 200g of fruits; 30g of nuts; and a cup of probiotic yogurt.
  Guided dietary follow-up was conducted through video viewing and WeChat or telephone follow-up. The researcher will provide cooking instruction or dietary pattern guidance by sending videos every two weeks.
  Arms: intervention group

SUMMARY:
The goal of this clinical trial is to conduct a dietary intervention targeting HIV-specific gut microbiota alterations for primary ASCVD prevention and evaluate its effectiveness in preventing borderline ASCVD risk among HIV-infected patients. The main questions it aims to answer are:

* Explore the pivotal role of the gut-heart axis in the causal relationship between HIV infection and atherosclerotic cardiovascular disease.
* Develop a targeted dietary intervention focusing on gut microbiota to prevent the borderline risk of atherosclerotic cardiovascular disease in HIV-infected patients.
* Evaluate the effectiveness of the gut microbiota-targeted dietary intervention in reducing atherosclerotic cardiovascular disease risk among HIV-infected patients, altering gut microbiota composition, improving risk factors of atherosclerotic cardiovascular disease, and alleviating prodromal symptoms associated with atherosclerotic cardiovascular disease.

Participants in the intervention group will receive the gut microbiota-targeted dietary intervention thrice weekly for 3 months, accompanied by bi-weekly health education videos for the same duration. Meanwhile, the control group will continue routine follow-up and health education practices. The intervention will span three months, followed by a three-month follow-up period. Data collection will occur at baseline, 3 months, and 6 months.

DETAILED DESCRIPTION:
Methods and data:

1. Mendelian randomization A two-step, two-sample mendelian randomization will be employed to investigate the potential mediating roles of gut microbiota in the causal relationship between HIV and atherosclerotic cardiovascular disease. Utilizing GWAS summary statistics from the Medical Research Council Integrative Epidemiology Unit OpenGWAS data and the MiBioGen study, we will conduct univariable mendelian randomization. The first step involves examining the causal pathway of HIV infection on gut microbiota (the coefficient=α), followed by elucidating the influence of gut microbiota on the development of atherosclerotic cardiovascular disease (the coefficient=β). The multiplication of these estimates (α*β) will delineate the mediation effects attributed to gut microbiota. Identification of specific gut microbiota exhibiting substantial mediation effects will guide the selection of our targeted intervention.
2. Systematic review To establish an empirical research foundation, a systematic review will synthesize evidence concerning the correlation between dietary patterns and gut microbiota, as well as the relationship between microbiota and atherosclerotic cardiovascular disease among people living with HIV. A thorough systematic search across database including PubMed/MEDLINE, MEDLINE (Ovid), Embase (Ovid), CINAHL (EBSCO), Web of Science, and China National Knowledge Infrastructure (CNKI). Articles meeting predefined inclusion and exclusion criteria will undergo rigorous extraction and summarization processes.
3. Intervention design and expert evaluation The intervention protocol will be formulated, drawing from the gut microbiota identified demonstrating significant mediation effects in the causal association between HIV infection and atherosclerotic cardiovascular disease, along with insights gleaned from the systematic review. Subsequently, multidisciplinary experts will be invited to evaluate the drafted protocol using the FAME (Feasibility, Appropriateness, Meaningfulness and Effectiveness) scale developed by the Joanna Briggs Institute.
4. Pragmatic randomized controlled trial We utilize a pragmatic randomized controlled trial design to evaluate the effectiveness of dietary intervention in real-world conditions, without strict control, thereby enhancing the generalizability and clinical applicability of our study findings. Participants at Shenzhen Third People's Hospital, exhibiting HIV with a borderline risk of atherosclerotic cardiovascular disease (5% to <7.5%) determined by the pooled cohort equation, will be enrolled. Upon providing informed consent, participants will undergo dynamic randomization into intervention and control groups, aiming for a 1:1 ratio while preserving maximum unpredictability. The intervention group will receive the gut microbiota-targeted dietary intervention thrice weekly for 3 months, accompanied by bi-weekly health education videos for the same duration. Meanwhile, the control group will continue routine follow-up and health education practices. The intervention will span three months, followed by a three-month follow-up period. Data collection will occur at baseline, 3 months, and 6 months. Primary outcomes will assess atherosclerotic cardiovascular disease risk via the pooled cohort equation and evaluate gut microbiota diversity and composition. Secondary outcomes will encompass biomarkers and predictors associated with atherosclerotic cardiovascular disease, as well as symptoms related to the condition.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-infected patients diagnosed according to the diagnostic criteria of China AIDS diagnosis and treatment guidelines (2021 edition);
2. Aged 18 years and above;
3. PCE predicted ASCVD risk of 5% - <7.5%;
4. Those with a predicted survival time of >1 year;
5. No plans to leave the depth in the next 3 months;
6. Voluntary participation in this study and signing the informed consent.

Exclusion Criteria:

1. Those with a past history of CVD;
2. Those with HIV-related neurocognitive disorders and various serious opportunistic infections;
3. Those with diabetes mellitus;
4. Known nut allergy;
5. Planning to become pregnant within 6 months;
6. Are on lipid-lowering therapy or using any interfering medications or diets;
7. Are participating in other HIV-related or dietary intervention-related scientific research programs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ASCVD risk estimated by the PCE | baseline, 3-month and 6-month
  Use the pooled cohort equation to estimate the participants' 10-year ASCVD risks
The composition of gut microbiota | baseline and 3-month
  Fecal samples will be collected from study participants, and the composition of gut microbiota will be analyzed using 16S rRNA technology. Diversity Analysis: Bacterial richness and phylogenetic diversity within samples will be assessed using Faith's Phylogenetic Diversity and richness metrics. Taxonomic Composition: Relative abundance of specific bacterial taxa will be determined through statistical analyses performed using phyloseq v. 1.26 and ggplot2 v. 3. Differential Abundance: A differential abundance analysis of Operational Taxonomic Units will be conducted. Beta Diversity: Differences in gut bacterial patterns among subjects consuming different diets will be evaluated using Bray Curtis dissimilarity, Weighted UniFrac, and Unweighted UniFrac metrics. Multivariate Analysis: Principal Coordinates Analysis will be performed to assess variations in the microbiome associated with dietary interventions.

SECONDARY OUTCOMES:
fasting blood lipids | baseline, 3-month and 6-month
  Fasting venous blood will be collected by venepuncture and centrifuged (4 C, 4000 rpm, 10 min) before plasma and erythrocytes are separately aliquoted and frozen at -20 ℃ and then stored at -80 ℃. Automated biochemical analyzer will be used to test the HDL-C (mmol/L), LDL-C (mmol/L), TG (mmol/L), and TC (mmol/L).
blood pressure | baseline, 3-month and 6-month
  To measure blood pressure using the Omron automatic blood pressure monitor, first ensure the patient is relaxed and seated comfortably with their back supported and feet flat on the floor. Place the cuff around the upper arm at heart level, ensuring a snug fit without being too tight. Use the device's inflation bulb to gradually inflate the cuff until it's sufficiently tight to stop blood flow, then slowly deflate the cuff while listening for the heartbeat sounds using the device's sensor. Record the values displayed on the monitor for both systolic and diastolic pressures (mmHg). Repeat this process three times with a short rest period between each measurement, and calculate the average of the three readings for accurate results.
BMI | baseline, 3-month and 6-month
  To measure BMI (Body Mass Index), first, the individual's height and weight are required. The person should be barefoot and wearing light clothing. Using a calibrated scale, the person's weight is measured in kilograms (kg). Next, their height is measured in meters (m) using a stadiometer or similar device. To calculate BMI, the weight in kilograms is divided by the square of the height in meters (BMI = weight(kg) / height(m)^2).
ASCVD symptoms | baseline, 3-month and 6-month
  Use the ACS symptom checklist and Memorial symptom assessment scale-heart failure to estimate ASCVD-related symptoms. The ACS Symptom Checklist is a validated instrument comprising 13 items designed to assess symptoms associated with ACS. Participants are asked to indicate whether each symptom is present (1) or absent (0). Each symptom is analyzed individually, and there is no composite score. The Memorial Symptom Assessment Scale-Heart Failure comprises 32 items, categorized into three subscales: physiological symptoms (n=21), psychological symptoms (n=6), and heart failure symptoms (n=5). Symptoms are rated on presence, frequency, severity, and distress, with frequency, severity, and distress rated on a Likert scale of 1-4, where higher scores indicate higher frequency, severity or greater distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No